CLINICAL TRIAL: NCT03730987
Title: Hispanic Men Building Respect Education and Safety (Family Men) - Substudy Under Center for Latino Research Opportunities (CLaRO)
Brief Title: Hispanic Men Building Respect Education and Safety/ HoMBRES Manteniendo Respeto, Educacion y Seguridad.
Acronym: HoMBRES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Victoria Mitrani, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20170769; U54MD002266 (NIH)
Record Dates: First submitted 2018-10-16; First posted 2018-11-05 (Actual); Results first posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-09

CONDITIONS: Substance Abuse; Domestic Violence; HIV/AIDS
Keywords: Family Violence; Hispanic/Latino; Health Disparities; Migrant farmworkers
MeSH Terms: conditions — Substance-Related Disorders; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HoMBRES Intervention Group - Father (Experimental): Four sessions (2 sessions per week, approximately 1.5 hours each) with the fathers, in which facilitators conduct educational sessions; During the period of social distancing, interventions were remotely facilitated via a well-tested video platform accessible by a link sent to the participants' telephone, computer, tablet or IPad (approximately 1.5 hours each session. Intervention videos were followed up with a telephone call to respond to any questions participants may have had about the sessions and clarify (if needed) the material covered in the videos via telephone or videoconferences. Only fathers were included in this group.
  Interventions: Behavioral: HoMBReS intervention; Behavioral: Families Talking Together (FTT)
- Diabetes Prevention Intervention Group - Father (Active Comparator): One session of 1.5 hours held once per week. Session content will focus on the importance of physical activity, healthy eating, and maintaining a healthy weight. Only fathers were included in this group.
  Interventions: Behavioral: Diabetes Prevention Intervention
- HoMBRES Intervention Group - Adolescent (No Intervention): The adolescent received no intervention.
- Diabetes Prevention Intervention Group - Adolescent (No Intervention): The adolescent received no intervention.

INTERVENTIONS:
Behavioral: HoMBReS intervention — Adapted intervention based on social cognitive theory and empowerment education that aims to reduce risky sexual behaviors, substance abuse and HIV among recently immigrated rural and urban men.
  Other Names: HoMBReS
  Arms: HoMBRES Intervention Group - Father
Behavioral: Families Talking Together (FTT) — The brief intervention, is a parent-based intervention to teach parents effective strategies proven to reduce adolescent sexual risk behavior. The intervention specifically targets the parent (not the adolescent) to: promote communication skills, build parent-adolescent relationships, develop effective monitoring strategies, reduce alcohol use, risky sexual behaviors and prepare them to teach adolescents assertiveness and substance abuse refusal skills.
  Other Names: FTT
  Arms: HoMBRES Intervention Group - Father
Behavioral: Diabetes Prevention Intervention — Session content will focus on the importance of physical activity, healthy eating and maintaining a healthy weight.
  Arms: Diabetes Prevention Intervention Group - Father

SUMMARY:
The overall objective of this project is to adapt and enhance HoMBReS (Hispanic Men Building Respect, Education, and Safety within Families /Hombres Manteniendo Respeto, Educacion y Seguridad de Familia), a Center for Disease Control (CDC)-identified best-evidence HIV behavioral intervention designed to reduce substance abuse, family violence, and HIV/AIDS (SAVA) among sexually active heterosexual Latino seasonal farmworkers (LSFWs) in rural areas.

DETAILED DESCRIPTION:
The HoMBRES de Familia project study (HoMBRES) examined the efficacy of a culturally adapted group intervention program with fathers from a seasonal farm working community and an Urban community in South Florida. The HoMBRES intervention study adapted and tested the efficacy of an intervention that can be adopted, implemented, and sustained with Latino fathers who live or work in the farm industry, construction, services, self employed or any other work industry in the semi-rural areas and urban areas of Miami Dade County. The HoMBRES intervention seeked to reduce risk for the SAVA (Substance Abuse, Violence, and HIV/AIDS infection) syndemic among this group of men and their adolescent sons.

The intervention HoMBRES consisted of four sessions remotely facilitated via a well-tested video platform accessible by a link sent to the participants' telephone, computer, tablet or IPad (approximately 1.5 hours each session). Staff scheduled the times when participants will watch the videotaped sessions in order to be available for their questions. Intervention videos were followed up with a telephone call to discuss presentation and respond to any questions participants may have had about the sessions and clarify (if needed) the material covered in the videos via telephone. Video sessions were completed within two weeks time period. Participants in the control group received one single video on diabetes prevention. Both groups were followed up six months post baseline interview.

ELIGIBILITY:
Inclusion Criteria:

* male
* adults (age 18 or above)
* living in semirural and urban areas of Miami Dade
* Latino
* understand and speaks Spanish
* has an eligible son ( 11-17 years old)

Exclusion Criteria:

* father does not provide consent and permission for his son
* son does not provide assent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender identity is self-reported.
Enrollment: 244 (Actual)
Dates: Start 2019-04-19 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Behar-Zusman, PhD, Principal Investigator — University of Miami
Locations (1):
- Florida International University, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only the father received the study intervention and completed the questionnaires that were included in the data for the primary and secondary outcomes. The adolescent received no intervention.
Groups:
- HoMBRES Intervention Group - Father: Participants in the intervention study will receive the adapted HoMBRES intervention which consisted of four participatory lectures and discussion session with the facilitator. Only fathers participated in the intervention group.
- Diabetes Prevention Intervention Group - Father: Participants in the Diabetes group received a single participatory lecture on diabetes prevention and discussion session with the facilitator. Only Fathers participated in the Diabetes Prevention Intervention Group.
- HoMBRES Intervention Group - Adolescent: The adolescents with the fathers from the HIV/AIDS intervention did not receive any of the adult intervention sessions.
- Diabetes Prevention Intervention Group - Adolescent: The adolescent from the diabetes prevention intervention with the fathers did not receive the adult intervention.
Period: Overall Study
Arm/Group | HoMBRES Intervention Group - Father | Diabetes Prevention Intervention Group - Father | HoMBRES Intervention Group - Adolescent | Diabetes Prevention Intervention Group - Adolescent
Started | 61 | 61 | 61 | 61
Completed | 59 | 61 | 59 | 61
Not Completed | 2 | 0 | 2 | 0
Not completed — Lost to Follow-up | 2 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Only the father received the study intervention and completed the questionnaires that were included in the data for the primary outcomes. Youth were only included in the secondary outcomes. The adolescent received no intervention.
Groups:
- HoMBRES Intervention Group - Father: Participants in the intervention study will receive the adapted HoMBRES intervention which consisted of three participatory lectures and discussion session with the facilitator. Only fathers are included in this group.
- Diabetes Prevention Intervention Group - Father: Participants in the Diabetes group received a single participatory lecture on diabetes prevention and discussion session with the facilitator. Only fathers are included in this group.
- HoMBRES Intervention Group - Adolescent: Adolescent from the did not receive any intervention. They only participated in baseline and six months follow up.
- Diabetes Prevention Intervention Group - Adolescent: Adolescent did not receive any intervention. They only participated in baseline and six months follow up.
- Total: Total of all reporting groups
Arm/Group | HoMBRES Intervention Group - Father | Diabetes Prevention Intervention Group - Father | HoMBRES Intervention Group - Adolescent | Diabetes Prevention Intervention Group - Adolescent | Total
Number analyzed (Participants) | 61 | 61 | 61 | 61 | 244
Age, Continuous [Mean (Full Range); unit: years] | 42.5 [18 to 64] | 44.4 [18 to 66] | 13.9 [11 to 17] | 13.7 [11 to 17] | 28.6 [11 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 61 | 61 | 61 | 61 | 244
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 61 | 61 | 61 | 61 | 244
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Demographics data was collected from both Fathers and sons. Adolescents did not participate in the interventions sessions.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 9 | 5 | 5 | 8 | 27
    White | 33 | 46 | 51 | 44 | 174
    More than one race | 18 | 10 | 5 | 8 | 41
    Unknown or Not Reported | 1 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participant Fathers Self-reporting Engagement in Risky Sexual Behaviors
Description: The number of participants that responded 'yes' to any of the following questions on the PhenX Toolkit Sexual Risk Behavior will be reported as self-reporting engagement in risky sexual behaviors; a) engaging in unprotected sexual encounters, b) more than one partner, c) anal sex with man in the last 6 months.
Time Frame: At Baseline, at 6 months follow up
Population: Not all participants completed the questions required. Only the father received the study intervention and completed the questionnaires that were included in the data for the primary and secondary outcomes. The adolescent received no intervention and were not included in the dataset.
Measure: Count of Participants; unit: Participants
Groups:
- HoMBRES Intervention Group - Father: Participants in the intervention study will receive the adapted HoMBRES intervention which consisted of three participatory lectures and discussion session with the facilitator. Only fathers were included in this group.
- Diabetes Prevention Intervention Group - Father: Participants in the Diabetes group received a single participatory lecture on diabetes prevention and discussion session with the facilitator. Only fathers were included in this group.
Arm/Group | HoMBRES Intervention Group - Father | Diabetes Prevention Intervention Group - Father
Number analyzed (Participants) | 58 | 61
Participants
  Baseline: number analyzed (Participants) | 58 | 60
  Baseline | 42 | 38
  6 months follow up: number analyzed (Participants) | 55 | 61
  6 months follow up | 38 | 53

2. Primary Outcome: The Number of Participant Fathers Self-reporting Experiences of Intra-partner Violence
Description: As measured using the PhenX Toolkit Exposures to Violence self-reported instrument. The variable was recoded using four categories: (1) "Your partner physically hurt you; (2) Insult or talk down to you; (3) Threaten you with harm; (4) Scream or curse at you. The responses are scored on a Likert-type scale 1=Never, 2=Rarely, 3=Sometimes, 4=Frequently, and 5=Always. The number of participants reporting 3 or higher on the Likert scale to any of the four categories, will be recorded as experiencing intra-partner violence.
Time Frame: At Baseline, at 6 months
Population: Two participants did not complete the 6-months follow up interview in the HoMBRES group. Only the father received the study intervention and completed the questionnaires that were included in the data for the primary and secondary outcomes. The adolescent received no intervention and were not included in the dataset.
Measure: Count of Participants; unit: Participants
Groups:
- HoMBRES Intervention Group - Father: Participants in the intervention study will receive the adapted HoMBRES intervention which consisted of four participatory lectures and discussion session with the facilitator. Only fathers were included in this group.
Arm/Group | HoMBRES Intervention Group - Father | Diabetes Prevention Intervention Group - Father
Number analyzed (Participants) | 61 | 61
Participants
  Baseline | 10 | 9
  6 months follow up: number analyzed (Participants) | 59 | 61
  6 months follow up | 10 | 5

3. Primary Outcome: The Number of Days Participant Fathers Reported Drinking in the Past 90 Days.
Description: The number of days participant reported drinking in the past 90 days using the Time-Line Followback self-reported questionnaire.
Time Frame: At Baseline, at 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | HoMBRES Intervention Group - Father | Diabetes Prevention Intervention Group - Father
Number analyzed (Participants) | 61 | 61
days
  Baseline | 8.59 (15.26) | 6.72 (11.98)
  6 months follow up: number analyzed (Participants) | 59 | 61
  6 months follow up | 11.08 (20.20) | 8.48 (14.37)

4. Primary Outcome: HIV Knowledge as Measured by the Brief HIV Knowledge Questionnaire
Description: As measured by the Brief HIV Knowledge Questionnaire. The proportion of correct answers will be reported (ranging from 0 to 1), with a score closer to 1 indicating higher HIV knowledge.
Time Frame: At Baseline, at 6 months
Population: Two participants did not complete the 6-months follow up interview in the HoMBRES group. Only the father received the study intervention and completed the questionnaires that were included in the data for the primary outcomes and adolescents were only included in the secondary outcomes. The adolescent received no intervention and were not included in the primary outcome dataset.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HoMBRES Intervention Group - Father | Diabetes Prevention Intervention Group - Father
Number analyzed (Participants) | 61 | 61
units on a scale
  Baseline | 0.65 (0.18) | 0.65 (0.21)
  6-months follow up: number analyzed (Participants) | 59 | 61
  6-months follow up | 0.81 (0.19) | 0.69 (0.19)

5. Primary Outcome: HIV Self-Efficacy as Measured by Self-Efficacy for STI and HIV Scale
Description: Self-Efficacy for Sexually Transmitted Infection (STI) and HIV Scale is a 9-item scale measuring the level of confidence in the ability to prevent STI and HIV infection. The measure uses a 5-point Likert scale (1=not sure at all to 5= completely sure). Total score ranges 9 to 45, with a higher score indicating a higher level of HIV self-efficacy.
Time Frame: At Baseline, at 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HoMBRES Intervention Group - Father | Diabetes Prevention Intervention Group - Father
Number analyzed (Participants) | 61 | 61
score on a scale
  Baseline | 38.30 (5.10) | 38.80 (6.10)
  6 months follow up: number analyzed (Participants) | 59 | 61
  6 months follow up | 40.20 (3.70) | 38.50 (5.40)

6. Primary Outcome: The Number of Drinks Per Day Over the Past 90 Days.
Description: The number of drinks per day over the past 90 days using the Timeline Followback.
Time Frame: At Baseline, at 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: drinks per day
Arm/Group | HoMBRES Intervention Group - Father | Diabetes Prevention Intervention Group - Father
Number analyzed (Participants) | 61 | 61
drinks per day
  Baseline | 2.82 (3.15) | 2.35 (2.43)
  6 months follow up: number analyzed (Participants) | 59 | 61
  6 months follow up | 2.89 (3.23) | 3.06 (3.98)

7. Secondary Outcome: Level of Self-reported Communication With Son as Measured by the Parental Practicing Scale
Description: The self-reported Parenting Practices Scale has a total score ranging from 1-5, with higher scores indicating higher levels of parental monitoring among the fathers. The adolescents responded to the son's version of the scale.
Time Frame: At Baseline, At 6 months
Population: Two participants did not complete the 6-months follow up interview in the HoMBRES group. Only the father received the study intervention and completed the questionnaires that were included in the data for the primary and secondary outcomes. The adolescent did not receive any interventions and were not included in the dataset.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- HoMBRES Intervention Group - Adolescent: Adolescents from the Fathers' intervention group did not participate in the intervention sessions. They only participated in the baseline and follow up interviews.
- HoMBRES Diabetes Control Group - Adolescent: Adolescents from the Fathers' control group did not participate in the control group sessions. They only participated in the baseline and follow up interviews.
Arm/Group | HoMBRES Intervention Group - Father | Diabetes Prevention Intervention Group - Father | HoMBRES Intervention Group - Adolescent | HoMBRES Diabetes Control Group - Adolescent
Number analyzed (Participants) | 61 | 61 | 61 | 61
score on a scale
  Baseline | 4.1 (0.8) | 4.3 (0.6) | 3.41 (0.92) | 3.36 (0.96)
  6 months follow up: number analyzed (Participants) | 59 | 61 | 61 | 61
  6 months follow up | 4.2 (0.6) | 4.4 (0.6) | 3.27 (1.09) | 3.47 (1.07)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- HoMBRES Intervention Group - Father: Four sessions (2 sessions per week, approximately 1.5 hours each) with the fathers, in which facilitators conduct educational sessions with groups of 6-8 men per group. One of the sessions includes an intervention of families talking together. Only fathers were included in this group.
  HoMBReS intervention: The experimental group (group A) will receive an intervention based on social cognitive theory and empowerment education that aims to reduce risky sexual behaviors among recently migrated rural men.
  Families Talking Together (FTT): The brief intervention, is a parent-based intervention to teach parents effective strategies proven to reduce adolescent sexual risk behavior. The intervention specifically targets the parent (not the adolescent) to: promote communication skills, build parent-adolescent relationships, develop effective monitoring strategies, and prepare them to teach adolescents assertiveness and substance abuse refusal skills.
- HoMBRES Intervention Group - Adolescent; Diabetes Prevention Intervention Group - Adolescent: Adolescent did not received intervention. They only participated in the baseline and six month follow up interviews.
Arm/Group | HoMBRES Intervention Group - Father | Diabetes Prevention Intervention Group - Father | HoMBRES Intervention Group - Adolescent | Diabetes Prevention Intervention Group - Adolescent
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/61 | 0/61 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/61 | 0/61 | 0/61
Other Adverse Events (participants affected / at risk) | 0/61 | 0/61 | 0/61 | 0/61

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-12): https://cdn.clinicaltrials.gov/large-docs/87/NCT03730987/Prot_SAP_001.pdf
  • Informed Consent Form (2020-04-12): https://cdn.clinicaltrials.gov/large-docs/87/NCT03730987/ICF_000.pdf